CLINICAL TRIAL: NCT00379587
Title: A Phase II Trial of Prophylactic Rituximab Therapy for Prevention of Chronic Graft-vs.-Host Disease After Allogeneic Stem Cell Transplantation
Brief Title: Rituximab for Prevention of Chronic GVHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry); Biogen (Industry)
Responsible Party: Principal Investigator, Corey S. Cutler, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05-377
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Results first posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-02

CONDITIONS: Hematological Malignancies
Keywords: Rituximab; Chronic GVHD
MeSH Terms: conditions — Hematologic Neoplasms; Bronchiolitis Obliterans Syndrome | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab at months 3, 6, 9 and 12 post-transplant
Drug: 375 mg/m2 RRituximab — Rituximab 375 mg/m2 q3months

SUMMARY:
The purpose of this trial is to determine if administration of rituximab after allogeneic stem cell transplantation can reduce the incidence of chronic GVHD. Chronic GVHD is a medical condition that can occur after bone marrow or stem cells are transplanted form one individual to another. After the transplant, the donor immune system may recognize the recipient body as foreign and may attempt to "reject" the body. Rituximab is a drug that interferes with the immune system function by specifically targeting B cells and killing them.

DETAILED DESCRIPTION:
Study Design: The study is designed as a Phase II, open label trial of Rituximab as chronic GVHD prophylaxis after HLA-matched, related or unrelated peripheral blood stem cell transplantation after ablative or non-ablative conditioning.

Primary Objective: To determine the incidence of clinically extensive chronic GVHD at one and two years after allogeneic stem cell transplantation after a single dose of Rituximab administered at 100 days, 6 months, 9 months and 1 year from transplantation as chronic GVHD prophylaxis.

Secondary Objectives: To determine the incidence of adverse hematological events, the incidence of infectious complications, the rate of malignant relapse, and the effects on donor hematopoietic chimerism after Rituximab administration.

Eligibility Criteria: Eligible patients will be 18 years of age or greater and will have undergone a non-myeloablative or fully ablative transplantation from an HLA-matched (6/6 loci) or single antigen/allele mismatched (5/6) donor approximately 100 days ago. Adequate performance status and organ function will be confirmed prior to enrollment. No ongoing infection or acute GVHD will be present at the time of enrollment. Evidence of sustained donor chimerism will be confirmed prior to study entry.

Treatment Description: Chronic GVHD prophylaxis will consist of Rituximab 375 mg/m2 administered 100 days, 6, 9 and 12 months after transplantation.

Accrual Objective: 68 patients will be accrued over 12 months.

Study Duration: Patients will be evaluated for two years after the time of transplantation for evaluation of the primary and secondary endpoints. Subjects will be followed longitudinally after completion of the study period for determination of clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone either ablative or non-myeloablative allogeneic stem cell transplantation
* Peripheral blood stem cells must have been used as the stem cell source
* Patients must have received transplantation from donors who are identical at 6 HLA loci, or mismatched at no more than 1 locus.
* Patients who have undergone a non-myeloablative stem cell transplant must have > 80% donor hematopoiesis within 30 days of study enrollment
* 18 years of age or older
* Performance Status 0-2
* Life expectancy of > 100 days
* Subjects with CLL are eligible, if there is no more than 20% residual leukemia in the bone marrow at the time of study entry

Exclusion Criteria:

* Evidence of relapsed or residual malignancy within 30 days of trial entry
* Highly aggressive B cell malignancy, such as Burkitt's lymphoma or Burkitt's-like lymphoma
* Allogeneic stem cell transplantation using a single or multiple umbilical cord blood units or using bone marrow
* Evidence of any active uncontrolled infection, or evidence of natural exposure to Hepatitis B, Hepatitis C or HIV
* Evidence of ongoing gastrointestinal or hepatic acute GVHD, or evidence of greater than ongoing Stage I cutaneous acute GVHD
* GVHD with chronic features diagnosed prior to day +100 or prior to enrollment
* Participation in a clinical trial evaluating another preventative strategy for chronic GVHD, or ongoing participation in a clinical trial for therapy of acute GVHD
* No Donor Lymphocyte Infusion (DLI) prior to day 100 and not plans for a DLI in the upcoming 30 days
* Heart failure uncontrolled by medications
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Cutler, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Cutler C, Kim HT, Bindra B, Sarantopoulos S, Ho VT, Chen YB, Rosenblatt J, McDonough S, Watanaboonyongcharoen P, Armand P, Koreth J, Glotzbecker B, Alyea E, Blazar BR, Soiffer RJ, Ritz J, Antin JH. Rituximab prophylaxis prevents corticosteroid-requiring chronic GVHD after allogeneic peripheral blood stem cell transplantation: results of a phase 2 trial. Blood. 2013 Aug 22;122(8):1510-7. doi: 10.1182/blood-2013-04-495895. Epub 2013 Jul 16. PMID 23861248

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituxan (Rituximab): 375mg/m^2 IV at 3, 6, 9 and 12 months from transplantation
Period: Overall Study
Arm/Group | Rituxan (Rituximab)
Started | 65
Completed | 63
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rituxan (Rituximab)
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 54 [19 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Clinician-diagnosed Chronic GVHD at One and Two Years
Time Frame: by 1 and 2 years after peripheral blood stem cell (PBSC) infusion
Measure: Number; unit: percentage of participants
Arm/Group | Rituxan (Rituximab)
Number analyzed (Participants) | 65
percentage of participants
  Year One | 38
  Year Two | 48

2. Secondary Outcome: Incidence of Grade 3 or Higher Infectious Complications
Time Frame: by 1 and 2 years after peripheral blood stem cell (PBSC) infusion
Measure: Number; unit: percentage of participants
Arm/Group | Rituxan (Rituximab)
Number analyzed (Participants) | 65
percentage of participants
  Year One | 11
  Year Two | 15

3. Secondary Outcome: Incidence of Relapse or Progression of Disease
Description: Percentage of participants with relapsed disease by year 4 post transplant.
Time Frame: by 4 years after peripheral blood stem cell (PBSC) infusion
Measure: Number; unit: percentage of participants
Arm/Group | Rituxan (Rituximab)
Number analyzed (Participants) | 65
percentage of participants | 34

4. Secondary Outcome: Incidence of Adverse Hematological Events
Description: White blood cell decrease, neutrophil cell count decrease, or platelet cell decrease considered possibly or probably related to therapy with rituximab.
Time Frame: by 18 months after peripheral blood stem (PBSC) infusion
Measure: Number; unit: participants
Arm/Group | Rituxan (Rituximab)
Number analyzed (Participants) | 65
participants | 11

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) inlcude events starting on or after day 0 and on or before day 540.
Description: If a subject experienced more than 1 of a given AE, the subject is counted only once for that AE. If a subject experienced more than 1 AE in a system organ class (SOC), the subject is counted only once in that SOC.
Arm/Group | Rituxan (Rituximab)
Serious Adverse Events (participants affected / at risk) | 6/65
Other Adverse Events (participants affected / at risk) | 22/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituxan (Rituximab) (N=65)
Septic Shock (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Interstital Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituxan (Rituximab) (N=65)
Hemoglobin Decrease (Blood and lymphatic system disorders) | 4
Neutrophil Decrease (Blood and lymphatic system disorders) | 7
Platelet Decrease (Blood and lymphatic system disorders) | 4
Fatigue (General disorders) | 5
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 4
Mucositis (Gastrointestinal disorders) | 4
Alkaline Phosphatase Increase (Blood and lymphatic system disorders) | 4
Alanine Aminotransferase Increase (Blood and lymphatic system disorders) | 6
Aspartate Aminotransferase Increase (Blood and lymphatic system disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes